CLINICAL TRIAL: NCT03650998
Title: Ultrasound-guided Transmuscular Quadratus Lumborum Block for Laparoscopic Hysterectomy. A Double Blind, Randomized, Placebo Controlled Trial.
Brief Title: Transmuscular Quadratus Lumborum Block for Total Laparoscopic Hysterectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZUH-TQL-TLH
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Pain
Keywords: nerve block; ultrasound; opioids; hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Active bilateral ultrasound-guided transmuscular quadratus lumborum (TQL) block. 60 mL ropivacaine 0.375% single shot.
  In both arms morphine will be administered IV as part of a patient controlled analgesia PCA)-pump regimen or additionally after contact with the nursing staff as it is the standard treatment.
  Interventions: Drug: Ropivacaine
- Placebo (Placebo Comparator): Placebo bilateral ultrasound-guided transmuscular quadratus lumborum (TQL) block. 60 mL Saline single shot.
  In both arms morphine will be administered IV as part of a patient controlled analgesia PCA)-pump regimen or additionally after contact with the nursing staff as it is the standard treatment.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — See arm description
  Arms: Active
Drug: Saline — See arm description
  Arms: Placebo

SUMMARY:
Study is designed to assess the effect of the transmuscular quadratus lumborum block on postoperative opioid consumption and pain for patients undergoing laparoscopic hysterectomy. Study is randomized, placebo-controlled and blinded. Seventy patients will be included.

DETAILED DESCRIPTION:
Every year three hundred patients undergo hysterectomy at the department of obstetric and gynaecologic surgery at Zealand University Hospital, University of Copenhagen. The most common procedure is Total Laparoscopic Hysterectomy (TLH), which is the preferred technique in about four out of five hysterectomies at our facility. Multimodal analgesia consists of Paracetamol 1 g, Ibuprofen 400 mg and Dexamethasone 8 mg and Sufentanil 0.2 micrograms/kg for emergence if no contraindications are present. Standard general anaesthesia is total intravenous anaesthesia (TIVA) with an induction consisting of Remifentanil and Propofol infusions, a bolus of Propofol followed by muscle relaxation with Rocuronium. Patients are intubated in the trachea. Anaesthesia is maintained with Remifentanil and Propofol infusions and boluses of Rocuronium are administered whenever the surgeon requires it. Patients are always in Trendelenburg's position. Thirty minutes prior to emergence a bolus of Sufentanil 0.2 microg/kg is administered, as mentioned previously. Of interest: two other different opioid based regimens are currently used in the other two hospitals in Region Zealand where this procedure is performed. There is no national standards defined for dosages used for this kind of surgery. Additionally, no regional techniques are defined for this surgical procedure.

Our research group at Zealand University Hospital has conducted a thorough retrospective one-year survey for this patient group in order to define the quantity of the research problem. The electronic anaesthesia files, PACU files and ward files were meticulously reviewed. The survey revealed an accumulated morphine consumption in the first 12 postoperative hours of 44.1±30.8 mg of oral morphine equivalents in TLH patients. This dosage should be evaluated in relation to the standardized multimodal regimen described above.

Anaesthesiologists have primarily used either epidural catheters or long-lasting opioids as the basis for the postoperative pain management of expected or manifest moderate to severe pain. An epidural blockade can be contraindicated for some patients, and might cause bladder paralysis, lower extremity paralysis, hypotension etc. In addition, the epidural technique is labour-intensive in application as well as in its requirements for monitoring. Thus, the continuous epidural blockade is not a possibility of interest to the gynaecologists at our hospital. Therefore, until recently, opioids have been the sole treatment of pain, when over-the-counter medicine does not suffice. This presents a problem for the patients due to the well-known adverse effects of morphine including postoperative nausea and vomiting (PONV), itching, fatigue, constipation, confusion, respiratory depression and delayed mobilization.

Postoperative complications to surgery are more frequent in patients experiencing postoperative pain, and besides reducing the immediate postoperative pain perception, the investigators consider reduction of the total morphine consumption and the potential of reducing development of chronic pain through better treatment of the acute pain, as very interesting and promising for the patients in our study.

The investigators have the technical capability to improve perioperative pain management by taking advantage of USG peripheral nerve blocks (PNBs). The investigators' group of researchers have described the transmuscular quadratus lumborum (TQL) block and the mechanism by which the TQL block works has been proven in a major cadaveric study and some case reports.

The TQL block is applied with the patient in the lateral position, with the side to be blocked turned upwards. The ultrasound transducer is placed in the transverse position at the posterior axillary line, just above the iliac crest, and adjusted to visualize the QL and psoas major (PM) muscles and the transverse process of vertebrae L3 or L4. The needle is subsequently inserted at the posterolateral end of the transducer and advanced in plane. The needle is advanced through the QL muscle until the tip of the needle penetrates the investing fascia of the QL muscle. The local anaesthetic is then injected in the interfascial plane, but posterior to the transversalis fascia (TF) and between the QL and PM muscles. Confirmation of correct application can subsequently be visualized when the two muscles are seen to spread apart on the ultrasound image.

The investigators want to perform evidence-based research using the USG TQL for patients undergoing TLH. The hypothesis is that the USG TQL block administered bilaterally and applied pre-operatively in the PACU or in the theatre for the TLH patients can reduce the postoperative morphine consumption by 50 % during the first 12 postoperative hours. It is considered a block with very little discomfort for the patient.

All patients scheduled for a TLH will be screened according to the inclusion and exclusion criteria. The suitable candidates will be asked prior to surgery, whether they want to participate in the trial. If so, before elective TLH, the patient will receive the block, allocated in a randomised fashion to either active LA or placebo. The block will be performed under standard perioperative monitoring by a trained and skilled physician from the department of anaesthesia. The active treatment will be a bilateral TQL block with 30 mL Ropivacaine 0.375% on each side, whereas the placebo group will receive the same volume of isotonic Saline, applied in the exact same way. The patients will all receive the same multimodal analgesic regimens, consisting of 1 g Acetaminophen, 400 mg Ibuprofen and 8 mg of Dexamethasone prior to surgery, and a regimen of 3 x Ibuprofen and 4 x Acetaminophen a day until discharge. An IV Morphine Patient-Controlled Analgesia (PCA) - pump will be used for 24 hours after instructions are given and the pump is set to begin in the PACU. In order to keep the pooled administration of local anaesthetic below the accepted maximum recommended dosage, neither local anaesthetic infiltration performed by the surgeon nor supplemental rescue regional techniques will be performed. Whenever pain exceeds an NRS of three despite the primary use of the PCA pump, the PACU nurses will administer additional Morphine or Sufentanil as they already do by the present standards.

Aim:

The aim with this study is to investigate the efficacy of the USG TQL block vs. Placebo in patients undergoing TLH.

The hypothesis is that the bilateral TQL block will significantly reduce the opioid consumption during the first 12 postoperative hours and significantly reduce the Numerical Rating Scale (NRS) pain score (0-10/10) and opioid related side effects.

Outcome:

Primary outcome:

The primary outcome of the study will be:

Morphine consumption in the first 12 postoperative hours (data from PCA pump and the patient's medical record).

The secondary outcomes will be:

(A) Pain intensity (NRS 0-10/10) in the study period at T0 (arrival in the PACU), after 15, 30 and 45 minutes. And again at 1, 2, 3, 4, 5, 6, 8, 10, 12, 15, 18, 21 and 24 hours postoperatively. In addition, NRS score will be recorded electronically in relation to all morphine administrations, since all patients must enter their NRS pain score on the PCA pump display in relation to administration of the PCA boluses.

(B) Total morphine consumption. Morphine consumption at 3, 6, 9, 12, 18 and 24 postoperative hours.

(C) Duration of block (time to first opioid). (D) Patient satisfaction with application of the block. (E) The degree of morphine-related side effects (PONV, itching, fatigue, etc.). (F) Time from operation to ambulation. The investigators regard these outcome parameters as essential for the selected patient group, and it is the investigators' hope that this could lead to a better amelioration of postoperative pain and reduced morphine consumption postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for TLH
* Age ≥ 18 years at the date of inclusion Have received thorough information, orally and in written, and signed the "Informed Consent" form on participation in the trial

Exclusion Criteria:

* Inability to cooperate
* Inability to speak, read and understand Danish
* Allergy to local anaesthetics or opioids
* Daily intake of opioids, according to the investigators decision
* Local infection at the site of injection or systemic infection
* Difficulty visualisation of muscular and fascial structures in ultrasound visualisation necessary to the block administration
* Co-morbidity, ASA>3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Hysterectomy requires a uterus.
Enrollment: 70 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | Twelve hours postoperatively
  How much cumulated opioid in oral morphine equivalents does the participant require/use.

SECONDARY OUTCOMES:
Postoperative pain intensity | 12 hours.
  NRS scale of 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Borglum, Ph.D.; MD, Study Chair — Consultant, associate professor.
Locations (1):
- Zealand University Hospital, Department of Anaesthesiology, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen C, Dam M, Nielsen MV, Tanggaard KB, Poulsen TD, Bendtsen TF, Borglum J. Transmuscular quadratus lumborum block for total laparoscopic hysterectomy: a double-blind, randomized, placebo-controlled trial. Reg Anesth Pain Med. 2021 Jan;46(1):25-30. doi: 10.1136/rapm-2020-101931. Epub 2020 Oct 20. PMID 33082286